CLINICAL TRIAL: NCT01420224
Title: Study of the Effects of Commercial Air Travel on Pulmonary Artery Pressure in Healthy Passengers and in a Patient With Chuvash Polycythaemia
Brief Title: Study of the Effects of Commercial Air Travel on the Lungs
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Ms Heather House, Head of Clinical Trials and Research Governance, University of Oxford
Other Study IDs: Oxford in-flight 2011
Record Dates: First submitted 2011-08-18; First posted 2011-08-19 (Estimated); Last update posted 2011-08-19 (Estimated); Status verified 2011-08

CONDITIONS: Healthy Volunteers; Chuvash Polycythaemia
Keywords: Air travel; Aircraft cabin hypoxia; Pulmonary artery pressure; Hypoxic pulmonary vasoconstriction; Pulmonary hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy volunteers
  Interventions: Other: Commercial airline flight
- Chuvash polycythaemia
  Interventions: Other: Commercial airline flight

INTERVENTIONS:
Other: Commercial airline flight — Normal scheduled passenger flight

SUMMARY:
The study hypothesis is that commercial air travel causes an increase in the blood pressure in the lungs (pulmonary artery pressure) that can be clinically relevant. Portable echocardiography (heart ultrasound) now offers a non-invasive means of studying this in-flight.

DETAILED DESCRIPTION:
In a commercial airliner flying at high altitude, the reduced cabin air pressure means that all passengers are exposed to slightly lowered oxygen levels ('hypoxia') equivalent to an altitude of approximately 5,000 to 8,000 ft. Although mild, this hypoxia is sufficient to stimulate some of the body's protective responses (eg changes in breathing and in hormonal secretion) and can be dangerous for passengers with heart or lung disease, who must breathe supplementary oxygen in-flight or may even be prohibited from flying because of the risks of hypoxia.

It is well known that severe hypoxia results in constriction of blood vessels in the lungs (a phenomenon called hypoxic pulmonary vasoconstriction), which in turn causes an increase in the blood pressure in the lungs ('pulmonary arterial pressure'). Unlike other physiological responses to hypoxia, this is often harmful and frequently leads to pulmonary hypertension and right heart failure (eg in some lung diseases and at high altitude). Even a modest increase in pulmonary arterial pressure could be clinically important in some airline passengers with heart/lung disease, as it may exacerbate their condition. However, it is not known whether the mild hypoxia experienced in an aircraft cabin is able to cause an increase in pulmonary artery pressure. Limited evidence suggests that it might - for example, there have been reports of passengers acutely developing new right heart failure in-flight, and data from animal studies also support this possibility.

This study aims to establish the effect of mild aircraft cabin hypoxia on pulmonary arterial pressure in healthy passengers and also in a patient with Chuvash polycythaemia. In this rare genetic disease, cellular responses to hypoxia are 'switched on' to some extent even during normoxia, causing increased red blood cell production. Affected individuals usually present with symptoms of polycythaemia in early adulthood and are typically asymptomatic following treatment with therapeutic venesection. Importantly, affected individuals have exaggerated acute hypoxic pulmonary vasoconstriction which may place them at risk of pulmonary hypertensive responses during air travel.

ELIGIBILITY:
For healthy volunteers:

Inclusion Criteria:

* suitable for echocardiographic measurements
* in good health

Exclusion Criteria:

* any significant medical condition

For patient with Chuvash polycythaemia:

Inclusion Criteria:

* diagnosis of Chuvash polycythaemia
* suitable for echocardiographic measurements

Exclusion Criteria:

* any other significant medical condition
* pulmonary hypertension
* uncontrolled erythrocytosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient with Chuvash polycythaemia recruited from previous study participants with the disease.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2011-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Systolic pulmonary artery pressure | In-flight
  The primary outcome measure is the effect of commercial air travel on systolic pulmonary artery pressure assessed by in-flight portable Doppler echocardiography.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Smith, MBBS DPhil FRCA, Principal Investigator — University of Oxford
Locations (1):
- University of Oxford, Oxford, United Kingdom